CLINICAL TRIAL: NCT05949502
Title: Evaluation of Performance and Occlusal Wear of Low Shrinkage Giomer Compared to Nanohybrid Resin Composite in Proximal Restorations After Two Years: A Randomized Clinical Trial.
Brief Title: Evaluation of Performance and Occlusal Wear of Low Shrinkage Giomer Compared to Nanohybrid Resin Composite
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omar Osama Shaalan, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Low shrinkage giomer
Record Dates: First submitted 2023-06-24; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Caries Class II
Keywords: Low-shrinkage Giomer; Nano-hybrid composite; Revised FDI criteria
MeSH Terms: interventions — ENA-HRi nano-hybrid composite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low shrinkage giomer. (Experimental): Low-shrinkage bioactive material (giomer) will be applied according to the manufacturer's instructions. Centripetal technique will be performed to restore the proximal wall followed by oblique incrementation of approximately 2 mm thick composite resin. This will be followed by light curing of each increment for 40 seconds using light curing unit till the whole cavity is filled.
  Interventions: Drug: Beautifil II LS (Low-Shrinkage)
- Nano-hybrid resin composite (Active Comparator): Nano-hybrid resin composite will be applied according to the manufacturer's instructions. Centripetal technique will be performed to restore the proximal wall followed by oblique incrementation of approximately 2 mm thick composite resin. Composite increments will be adapted obliquely on each cusp. This will be followed by light curing for 40 seconds using light curing unit of each increment till the whole cavity is filled.
  Interventions: Drug: 3M Filtek Z250 XT Universal

INTERVENTIONS:
Drug: Beautifil II LS (Low-Shrinkage) — low shrinkage bioactive material Giomer
  Other Names: low shrinkage Giomer
  Arms: Low shrinkage giomer.
Drug: 3M Filtek Z250 XT Universal — Universal Nano-hybrid composite
  Other Names: Nano-hybrid composite
  Arms: Nano-hybrid resin composite

SUMMARY:
A clinical trial, comparing the clinical performance and occlusal wear resistance of two different restorative materials in restoring proximal caries in permanent posterior teeth. One is based on giomer technology and the other is nano-hybrid resin composite.

DETAILED DESCRIPTION:
The aim of this study is to assess clinical performance and occlusal wear resistance of low shrinkage Giomer and Nanohybrid Resin Composite in proximal restorations using revised FDI (World Dental Federation) criteria and digital intra-oral scanner.

Two different restorative materials will be evaluated after two years for fracture, retention and occlusal wear. Furthermore, the rest of the revised FDI Criteria including functional (marginal adaptation, proximal contact point, form and contour, occlusion and occlusal wear) , biological (caries at restoration margin (CAR), dental hard tissue defects at restoration margin and postoperative hypersensitivity/pulp status) and esthetic properties (surface luster and surface texture, marginal staining and color match) will be also evaluated.

The first material is based on the giomer technology which is a true hybrid between nano-hybrid resin composite and glass ionomer. The comparator will be a nano-hybrid resin composite.

Examination and selection of all patients will be done. Teeth with proximal, primary carious lesions will be selected. Rubber dam isolation will be done followed by preparation of Class II cavities and placement of restorative material according to the randomization sequence.

Low-shrinkage bioactive material will be applied according to the manufacturer's instructions. For the comparator group, nano-hybrid resin composite will be also applied according to the manufacturer's instructions. Restorations will evaluated at baseline, after six, 12, 18 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for patients

  * Patient's age ranging from 19-30
  * Good oral hygiene.
  * Patients who have stable occlusion.
  * Patients who could be present for further periodic follow-ups.
  * Possibility for application of rubber dam during restoration.
  * Patient compliance.
* Inclusion criteria for Teeth

  * Vital first and second molars, with compound Class II lesions.
  * The selected teeth should be in occlusion with natural dentition and having proximal contact with adjacent teeth.
  * Healthy periodontium.

Exclusion Criteria:

* Exclusion criteria for patients

  * Poor oral hygiene.
  * Patients with high caries index or high plaque index.
  * Patients with periodontal problems.
  * Heavy bruxism habit or presence of any parafunctional habits.
  * Any allergic reactions against any components of the materials to be used in the study.
  * History of severe medical complications such as xerostomia.
  * Pregnant or lactating women.
  * Participating in another clinical trial.
* Exclusion criteria for teeth

  * Fractured or evidently cracked teeth.
  * Defective restorations adjacent or opposite the selected tooth for research.
  * Atypical extrinsic staining of teeth.
  * Teeth with defects or lesions requiring other operative interventions.
  * Teeth with pulpal pain.
  * Teeth with periapical lesions.
  * Root Canal treated teeth.
  * Mobile Teeth.
  * Non-functioning teeth with no opposing tooth.
  * Signs of severe attrition.
  * Heavy occlusion.
  * Periodontally affected teeth.

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Functional properties (F1) Fracture of material and retention according to revised FDI (World Dental Federation) criteria. Measured by visual examination and short air drying. | 24 months
  Method of aggregation is frequency and percentage. Measuring unit is scoring system (Ordinal, scores 1-5). (1) Clinically excellent. (sufficient). (5) Clinically poor (entirely insufficient).

SECONDARY OUTCOMES:
Quantitative occlusal restoration wear by Digital Intra-oral scanner and Geometrical subtraction software. | 24 months.
  Method of aggregation is Mean (SD) (parametric) or Median (Range) (Non-parametric). Measuring unit is Microns.
Functional properties according to revised FDI (World Dental Federation) criteria. | 24 months.
  Functional properties:
  F2: Marginal adaptation measured by visual examination, short air drying, 250 μm probe.
  F3:Proximal contact point measured by visual examination and 25/50/100 μm blades.
  F4: Form and contour measured by visual examination. F5: Occlusion and occlusal wear measured by visual examination and articulation paper.
  Method of aggregation is frequency and percentage. Measuring unit is scoring system (Ordinal, scores 1-5). (1) Clinically excellent. (sufficient). (5) Clinically poor (entirely insufficient).
Biological properties according to revised FDI criteria. | 24 months.
  Biological properties:
  B1: Caries at restoration margin (CAR) measured by visual examination, short air drying, and 250 μm probe.
  B2: Dental hard tissue defects at restoration margin measured by visual examination.
  B3: Postoperative hypersensitivity reported by patient and pulp status tested with cold stimulus.
  Method of aggregation is frequency and percentage. Measuring unit is scoring system (Ordinal, scores 1-5). (1) Clinically excellent. (sufficient). (5) Clinically poor (entirely insufficient).
Aesthetic properties according to revised FDI criteria. | 24 months.
  Aesthetic properties:
  A1: Surface luster and surface texture measured by visual examination and short air drying.
  A2: Marginal staining measured by visual examination and short air drying. A3: color match measured by visual examination. Method of aggregation is frequency and percentage. Measuring unit is scoring system (Ordinal, scores 1-5). (1) Clinically excellent. (sufficient). (5) Clinically poor (entirely insufficient).

IPD SHARING:
Plan to Share IPD: No